CLINICAL TRIAL: NCT05474118
Title: Real-life Use of Cefazolin for the Treatment of Meticillin-susceptible Staphylococcal Infective Endocarditis: Comparison to a Treatment Cohort With Penicillin M
Acronym: CEFASTA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 18-45b
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2021-09

CONDITIONS: Infectious Disease; Endocarditis
Keywords: cefazolin
MeSH Terms: conditions — Communicable Diseases; Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective, regional, multicenter study (including the Annecy-Genevois Hospital Center, the Chambéry Métropole Savoie Hospital Center, and the Grenoble University Hospital Center), comparing a cohort of patients treated with Cefazolin with a cohort of patients treated with Penicillin M

DETAILED DESCRIPTION:
The use of Cefazolin for the treatment of infective endocarditis caused by Staphylococcus meti - S has become commonplace in France following the stockout of injectable Penicillin M, the reference treatment, which occurred during 2016.

There is currently no clinical data to prejudge the efficacy of Cefazolin in the context of high inoculum, such as in the treatment of infective endocarditis.

On the other hand, recent data have described a better tolerance profile for Cefazolin than for Penicillin M.

The objective of this study is to compare the efficacy and safety of Cefazolin with that of Penicillin M in the management of methicillin-susceptible staphylococcal endocarditis, through the analysis of two retrospective cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Definite infective endocarditis according to Duke criteria
* Documented SAMS or meticillin-sensitive SCN
* Treated with Cefazolin or Penicillin M for at least 10 consecutive days
* Treatment initiated between 01/01/2014 and 12/31/2018

Exclusion Criteria:

* Patients under 18 years old
* Patients under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study are adults older than 18 years of age, who were treated between 01/01/2014 and 12/31/2018 for definite infective endocarditis according to Duke criteria. The infection must have been documented with Staphylococcus Meti -S, on native valve or device, and treated with Cefazolin or Penicillin M for at least 10 consecutive days.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficacy of Cefazolin in the treatment of Staphylococcus meti -S infective endocarditis, with that of Penicillin M, by observing the rate of death, relapse of infective endocarditis and occurence of embolic event. | Day 10 (End of antibiotic treatment according to national recommendations
  The primary outcome is management failure, a composite outcome defined by the existence of at least one of the following:
  * Death before the end of treatment
  * Relapse of infective endocarditis, with the same germ, within 3 months of the end of antibiotic therapy
  * Occurrence of embolic event after antibiotic therapy

SECONDARY OUTCOMES:
Assessment of clinical and biological tolerance | 10 days (Occurrence of adverse events during the antibiotic treatment period)
  Occurrence of adverse events such as: acute renal failure, coagulation disorder, cytolysis
Description of clinical predictive factors of failure | 10 days (during the antibiotic treatment period)
  Collection of clinical data in order to identify certain predictive factors of failure using directed acyclic graph.
Description of microbiological predictive factors of failure | 10 days (during the antibiotic treatment period)
  Collection of microbiological data in order to identify certain predictive factors of failure using directed acyclic graph.
Description of ultrasound predictive factors of failure | 10 days (during the antibiotic treatment period)
  Collection of ultrasound data in order to identify certain predictive factors of failure using directed acyclic graph.

CONTACTS AND LOCATIONS:
Overall Officials: Mylène Maillet, Principal Investigator — CH Annecy Genevois
Locations (1):
- Centre Hospitalier Annecy Genevois, Metz-Tessy, France